CLINICAL TRIAL: NCT06454058
Title: Association Between Euploid Embryo Grade and Maternal Age, a Retrospective Cross-sectional Study
Brief Title: Association Between Euploid Embryo Grade and Maternal Age
Status: Terminated | Type: Observational
Why Stopped: Preliminary findings of inconsistent embryo grading across sites.
Sponsor: Inception Fertility Research Institute, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: INC-IIS-2024-004
Record Dates: First submitted 2024-06-06; First posted 2024-06-12 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Fertility
Keywords: Advanced Maternal Age; Embryo Grade

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Background: Advanced maternal age (AMA) is associated with a reduction in live birth rate (LBR) after ART cycles. The main reason for this reduction is the lower number of oocytes aspirated, the number of developing embryos and the low number of euploid embryos available for transfer. The impact of age on success rates after the transfer of an euploid embryo has been a matter of discussion, with a recent meta-analysis showing a reduction in LBR after the transfer of an euploid blastocyst to women of AMA (1). There could be many reasons for this reduced LBR but they can be categorized into two broad categories - the uterus (including the mother's health) and the embryo (including the oocyte and the sperm).

It is possible that factors associated with reduced embryo quality would manifest in a lower embryo grade.

DETAILED DESCRIPTION:
Objective: To study if there is an association between advanced maternal age and lower embryo grading of euploid embryos.

Hypothesis: Advanced maternal age is associated with a lower embryonic grade in euploid embryos.

Study Design: This is a retrospective cross-sectional study of euploid embryos from patients who have completed IVF with PGT-A testing at a fertility clinic in The Prelude Network (US sites only). A comparison of embryo grade between different age groups (<35, 40+) will be done after controlling for baseline demographic characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have completed IVF egg retrieval with PGT-A testing at a fertility clinic in The Prelude Network (US clinics, excluding NYU)
* PGT biopsy was conducted in 2023,
* PGT biopsy was performed on blastocyst stage embryo,
* PGT-A result is euploid.

Exclusion Criteria:

* PGT-A result is mosaic,
* Embryos in which PGT-M was done and were found to be carriers of the mutation,
* Embryos in which PGT-SR was done and were found to be carriers of the structural rearrangement.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who have completed IVF egg retrieval with PGT-A testing at a fertility clinic in The Prelude Network (US clinics, excluding NYU).
Sampling Method: Non-Probability Sample
Enrollment: 502 (Actual)
Dates: Start 2024-06-07 (Actual); Primary Completion 2025-03-26 (Actual); Study Completion 2025-03-26 (Actual)

PRIMARY OUTCOMES:
Embryo Grade | 6 months
  Embryo grade for PGT-A confirmed euploid embryos

CONTACTS AND LOCATIONS:
Locations (1):
- Inception Fertility Research Institute, LLC, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vitagliano A, Paffoni A, Vigano P. Does maternal age affect assisted reproduction technology success rates after euploid embryo transfer? A systematic review and meta-analysis. Fertil Steril. 2023 Aug;120(2):251-265. doi: 10.1016/j.fertnstert.2023.02.036. Epub 2023 Mar 5. PMID 36878347